CLINICAL TRIAL: NCT04603066
Title: Administration of Ondansetron With P-glycoprotein Inhibitor Tariquidar in Patients With Neuropathic Pain
Brief Title: Tariquidar-ondansetron Combination in Neuropathic Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, simon.haroutounian, Associate Professor, Washington University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 202008183
Record Dates: First submitted 2020-09-21; First posted 2020-10-26 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Ondansetron; tariquidar

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double blind, crossover study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ondansetron/Placebo first, then Ondansetron/Tariquidar (Other): The study group where patients received Ondansetron with Placebo during Visit 1, and after a washout period of 3 weeks Ondansetron with Tariquidar at Visit 2 per the randomization schedule.
  Ondansetron 16 mg was administered IV over 60 minutes with placebo (D5W) or with tariquidar (4mg/kg dose in D5W). Ondansetron was diluted in 100mL 0.9% normal saline, and tariquidar was diluted in 500mL D5W.
  Interventions: Drug: Ondansetron 16 mg with Tariquidar; Drug: Ondansetron 16 mg with Placebo
- Ondansetron/Tariquidar first, then Ondansetron/Placebo (Other): The study group where patients received Ondansetron with Tariquidar during Visit 1, and after 3 weeks of washout period Ondansetron with Placebo at Visit 2 per the randomization schedule.
  Ondansetron 16 mg was administered IV over 60 minutes with tariquidar (4mg/kg dose in D5W) or with placebo (D5W). Ondansetron was diluted in 100mL 0.9% normal saline, and tariquidar was diluted in 500mL D5W.
  Interventions: Drug: Ondansetron 16 mg with Tariquidar; Drug: Ondansetron 16 mg with Placebo

INTERVENTIONS:
Drug: Ondansetron 16 mg with Tariquidar — In randomized order, each participant will receive two IV infusions of ondansetron, 3 weeks apart; one with placebo (D5W), and one with tariquidar (4mg/kg dose in D5W) administered IV over 60 minutes. Ondansetron will be diluted in 100mL 0.9% normal saline, and tariquidar will be diluted in 500mL D5W.
  Other Names: Ondansetron/Tariquidar
Drug: Ondansetron 16 mg with Placebo — In randomized order, each participant will receive two IV infusions of ondansetron, 3 weeks apart; one with placebo (D5W), and one with tariquidar (4mg/kg dose in D5W) administered IV over 60 minutes. Ondansetron will be diluted in 100mL 0.9% normal saline, and tariquidar will be diluted in 500mL D5W.
  Other Names: Ondansetron/ Placebo

SUMMARY:
Prospective, randomized, double-blind, placebo controlled, cross-over proof of concept study.

To determine the pharmacokinetics and tolerability of co-administration of 5-HT3R antagonist ondansetron with a P-glycoprotein inhibitor tariquidar, in patients with neuropathic pain.

DETAILED DESCRIPTION:
The investigators hypothesize that co-administration of a 5-HT3 receptor antagonist ondansetron (single 16mg dose) with p-glycoprotein inhibitor tariquidar (single 4mg/kg dose) vs placebo in a cross-over prospective randomized study, will:

1. Be tolerable in patients with neuropathic pain.
2. Increase the cerebrospinal fluid (CSF) to plasma ratio of ondansetron after intravenous administration, compare to ondansetron alone
3. Result in a greater reduction in pain intensity than with ondansetron alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65;
2. Documented diagnosis of neuropathic pain due to damage or disease affecting the peripheral nervous system;
3. At least Probable neuropathic pain grading1;
4. Pain duration >3 months;
5. Average pain intensity ≥4 on 0-10 numerical rating scale (NRS).

Exclusion Criteria:

1. Current pregnancy or lactation;
2. Moderate-severe kidney or liver dysfunction;
3. Active cardiac arrhythmias (non-sinus rhythm), Long QT syndrome, or QTc interval >450msec;
4. Congestive heart failure
5. Abnormal troponin values at screening visit;
6. Current treatment with MAO inhibitors, mirtazapine, SSRI antidepressants, or SNRI medications duloxetine or venlafaxine;
7. Current treatment with tapentadol, tramadol, or fentanyl;
8. Current treatment with P-glycoprotein substrate drugs with narrow therapeutic window, e.g. digoxin;
9. Current treatment with tricyclic antidepressant medications (e.g. amitriptyline, desipramine, imipramine) at a dose >25mg/day;
10. Ongoing use of any of the following medications with known effects on Pgp function: carbamazepine, phenytoin, phenobarbital, cyclosporine, clarithromycin, erythromycin, ritonavir, verapamil, rifampicin, St. John's wort;
11. Current treatment with QT-prolonging drugs, and drugs known to have a significant interaction with ondansetron or other P-glycoprotein substrates (see section 2.3.3.);
12. Current treatment with anticoagulant drugs;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-31 (Actual); Primary Completion 2023-10-21 (Actual); Study Completion 2023-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Haroutounian, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine/Barnes-Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Finnerup NB, Haroutounian S, Kamerman P, Baron R, Bennett DLH, Bouhassira D, Cruccu G, Freeman R, Hansson P, Nurmikko T, Raja SN, Rice ASC, Serra J, Smith BH, Treede RD, Jensen TS. Neuropathic pain: an updated grading system for research and clinical practice. Pain. 2016 Aug;157(8):1599-1606. doi: 10.1097/j.pain.0000000000000492. PMID 27115670
- [Background] Yawn BP, Wollan PC, Weingarten TN, Watson JC, Hooten WM, Melton LJ 3rd. The prevalence of neuropathic pain: clinical evaluation compared with screening tools in a community population. Pain Med. 2009 Apr;10(3):586-93. doi: 10.1111/j.1526-4637.2009.00588.x. Epub 2009 Mar 17. PMID 20849570
- [Background] Smith BH, Torrance N. Epidemiology of neuropathic pain and its impact on quality of life. Curr Pain Headache Rep. 2012 Jun;16(3):191-8. doi: 10.1007/s11916-012-0256-0. PMID 22395856

RESULTS

PARTICIPANT FLOW:
Groups:
- Ondansetron/Placebo First, Then Ondasetron/Tariquidar: The study group where patients received Ondansetron with Placebo during Visit 1, and after a washout period of 3 weeks Ondansetron with Tariquidar at Visit 2 per the randomization schedule.
  Ondansetron 16 mg was administered IV over 60 minutes with placebo (D5W) or with tariquidar (4mg/kg dose in D5W). Ondansetron was diluted in 100mL 0.9% normal saline, and tariquidar was diluted in 500mL D5W.
Period: Visit 1
Arm/Group | Ondansetron/Placebo First, Then Ondasetron/Tariquidar | Ondansetron/Tariquidar First, Then Ondansetron/Placebo
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Wash-out (3 Weeks)
Arm/Group | Ondansetron/Placebo First, Then Ondasetron/Tariquidar | Ondansetron/Tariquidar First, Then Ondansetron/Placebo
Started | 12 | 12
Completed | 11 | 12
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0
Period: Visit 2
Arm/Group | Ondansetron/Placebo First, Then Ondasetron/Tariquidar | Ondansetron/Tariquidar First, Then Ondansetron/Placebo
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data from 24 enrolled patients were used in baseline analysis.
Groups:
- Ondansetron With Tariquidar First, Then Ondansetron With Placebo: The study group where patients received Ondansetron with Tariquidar during Visit 1, and Ondansetron with Placebo at Visit 2 per the randomization schedule. The washout period between two visits was 3 weeks.
  Ondansetron 16 mg was administered IV over 60 minutes with tariquidar (4mg/kg dose in D5W) or with placebo (D5W). Ondansetron was diluted in 100mL 0.9% normal saline, and tariquidar was diluted in 500mL D5W.
- Ondansetron With Placebo First, Then Ondansetron With Tariquidar: The study group where patients received Ondansetron with Placebo during Visit 1, and Ondansetron with Tariquidar at Visit 2 per the randomization schedule. The washout period between two visits was 3 weeks.
  Ondansetron 16 mg was administered IV over 60 minutes with placebo (D5W) or with tariquidar (4mg/kg dose in D5W). Ondansetron was diluted in 100mL 0.9% normal saline, and tariquidar was diluted in 500mL D5W.
- Total: Total of all reporting groups
Arm/Group | Ondansetron With Tariquidar First, Then Ondansetron With Placebo | Ondansetron With Placebo First, Then Ondansetron With Tariquidar | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (12.87) | 49.33 (12.16) | 50.92 (12.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 12 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Concertation-time Profile of Ondansetron in Plasma, Measured by the Area Under the Concentration-time Curve (AUC)
Description: AUCinf for Ondansetron concentration in plasma based on venous blood sampling for plasma concentrations of ondansetron obtained at 0, 15, 30, 60, 90, 120, 180, and 240 minutes from the beginning of ondansetron infusion.
Time Frame: Measurements over 240 minutes, extrapolated to infinity
Population: participants who completed both sessions
Measure: Mean (Standard Deviation); unit: mg*hr/L
Groups:
- Ondansetron + Tariquidar: Ondansetron 16 mg with Tariquidar: In randomized order, each participant will receive two IV infusions of ondansetron, 3 weeks apart; one with placebo (D5W), and one with tariquidar (4mg/kg dose in D5W) administered IV over 60 minutes. Ondansetron will be diluted in 100mL 0.9% normal saline, and tariquidar will be diluted in 500mL D5W.
- Ondansetron + Placebo: Ondansetron 16 mg with Placebo: In randomized order, each participant will receive two IV infusions of ondansetron, 3 weeks apart; one with placebo (D5W), and one with tariquidar (4mg/kg dose in D5W) administered IV over 60 minutes. Ondansetron will be diluted in 100mL 0.9% normal saline, and tariquidar will be diluted in 500mL D5W.
Arm/Group | Ondansetron + Tariquidar | Ondansetron + Placebo
Number analyzed (Participants) | 22 | 22
mg*hr/L | 0.89 (0.29) | 0.87 (0.45)
Statistical Analysis 1: Comparison: Ondansetron + Tariquidar vs Ondansetron + Placebo; Test type: Superiority; p = 0.8651, t-test, 2 sided; Mean Difference (Final Values) = 0.0204257, 95% CI 2-sided [-0.2624635 to 0.2216122]

2. Primary Outcome: Cerebrospinal Fluid to Plasma Concentration Ratio of Ondansetron
Description: The level of ondansetron in plasma and CSF (cerebrospinal fluid) in samples, taken around the same time, was measured, and the ratio of the two values was calculated. This ratio (partition coefficient, Kp) of ondansetron, compared between the two sessions, with placebo vs tariquidar
Time Frame: anytime between 0-240 minutes
Population: Participant who had both CSF and plasma samples drawn at the same time, at both sessions.
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Ondansetron + Tariquidar | Ondansetron + Placebo
Number analyzed (Participants) | 7 | 7
ratio | 0.132 (0.017) | 0.112 (0.018)
Statistical Analysis 1: Comparison: Ondansetron + Tariquidar vs Ondansetron + Placebo; Test type: Superiority; p = 0.056, t-test, 2 sided; Mean Difference (Net) = 0.01727052, 95% CI 2-sided [-0.0005895 to 0.03513063]

3. Secondary Outcome: % Change in Pain Intensity
Description: Change in spontaneous pain intensity (measured on a 0-10 numerical rating scale; 0=no pain, 10=worst imaginable pain) from baseline to 90 minutes after ondansetron IV infusion, compared between two sessions with and without tariquidar. Values are presented as a percentage change from baseline.
Time Frame: baseline to 90 minutes after ondansetron IV infusion
Population: All patients who received both treatments, excluding pharmacokinetic outlier (patient N 06)
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | Ondansetron + Tariquidar | Ondansetron + Placebo
Number analyzed (Participants) | 22 | 22
% change from baseline | 37.2 (35.1) | 28.8 (28.7)

4. Secondary Outcome: Conditioned Pain Modulation (CPM) Magnitude (ΔCPM)
Description: Conditioned Pain Modulation (CPM) is a psychophysical test to assess the efficiency of descending pain inhibition. CPM is calculated as difference in heat pain threshold with and without pain conditioning - i.e. immersion of a hand in cold water. Conditioned Pain Modulation (CPM) Negative CPM values represent efficient pain modulation/inhibition.
  This test was administered at baseline, and again 90-min after the end of ondansetron infusion. CPM values can range from -100 to 100, CPM<0 (i.e. decreased pain to heat stimulus following conditioning) implies descending pain inhibition.
  CPM Magnitude (ΔCPM) is the calculated by subtracting the measurement of CPM at baseline [possible range of CPM scores 0-100] from the measurement of CPM 90 min after the intervention [possible range of CPM scores 0-100]. A larger negative ΔCPM value indicates increased pain modulation efficiency following treatment, and therefore, a desired outcome.
Time Frame: Baseline and 90 minutes after the end of ondansetron infusion
Population: All patients who completed both CPM procedures
Measure: Mean (Standard Error); unit: score on a scale of 0-100
Arm/Group | Ondansetron + Tariquidar | Ondansetron + Placebo
Number analyzed (Participants) | 20 | 20
score on a scale of 0-100 | 0.1 (8.2) | 1.8 (10.4)

5. Secondary Outcome: Correlation Between CPM Magnitude (ΔCPM) and Change in Pain Intensity
Description: The association between baseline Conditioned Pain Modulation (CPM) magnitude (ΔCPM) and the % pain reduction from baseline will be determined by bivariate regression.
Time Frame: 0-240 min from infusion
Population: All patients who completed CPM and reported spontaneous pain intensity at corresponding time points
Measure: Number; unit: r2
Arm/Group | Ondansetron + Tariquidar | Ondansetron + Placebo
Number analyzed (Participants) | 20 | 20
r2 | 0.02 | 0.01

6. Secondary Outcome: Change in Neuropathic Pain Symptom Inventory (NPSI) Score
Description: Changes in the Neuropathic Pain Symptom Inventory (NPSI) total score will be compared between treatment sessions.
  NPSI is a questionnaire used to assess and quantify neuropathic pain by asking patients to rate the severity of different pain sensations on a scale of 0 to 10, with 0 being no pain and 10 being the worst pain imaginable. The version administered in the study consists of seven questions, each rated on a scale from 0 to 10, with the total score being the sum of all ratings.
  The possible range of the NPSI score of the version administered in the study is 70, and, since we measure the difference in scores, the changes in the NPSI score of the version administered in the study is -70 to 70. Higher NPSI scores indicate more severe neuropathic pain symptoms. Since the analysis is conducted on changes in NPSI scores from baseline, a more negative value corresponds to a greater reduction in neuropathic pain symptoms following treatment.
Time Frame: baseline to 70 min after infusion
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Ondansetron + Tariquidar | Ondansetron + Placebo
Number analyzed (Participants) | 22 | 22
units on a scale | -8.6 (7.0) | -13.2 (7.1)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Ondansetron + Tariquidar | Ondansetron + Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 12/23 | 19/24
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ondansetron + Tariquidar (N=23) | Ondansetron + Placebo (N=24)
Headache (Nervous system disorders) | 7 (7) | 7 (7)
Metallic Taste (Gastrointestinal disorders) | 8 (8) | 2 (2) — Dysgeusia (Change in taste)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Drowsiness (Nervous system disorders) | 7 (7) | 2 (2)
Nausea (Nervous system disorders) | 3 (3) | 5 (5)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 2 (2) | 2 (2) — specifically facial tingling
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 3 (3) | 0 (0) — Vasovagal response (syncope) during needle placement
Infusion site bruising (Skin and subcutaneous tissue disorders) | 8 (8) | 0 (0) — Pain/bruising/burning at infusion site

LIMITATIONS AND CAVEATS:
Due to ethical considerations, cerebrospinal fluid (CSF) sampling was optional in the study, therefore data on plasma/CSF ratio is not available for all patients.

A total of 24 patients were enrolled out of 28 participant planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT04603066/Prot_SAP_000.pdf